CLINICAL TRIAL: NCT01522339
Title: Pilot Study: Safety of a Customized MRI System for Neonatal Imaging
Acronym: NICU MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-2045
Record Dates: First submitted 2011-11-22; First posted 2012-01-31 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Safety of a Customized NICU MRI System
Keywords: NICU; MRI; Neonatal; Safety; Efficacy; Cincinnati

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Safety of a Customized NICU MRI System (Experimental): Device: GE OPTIMA MR430s with HDX/GE Electronics
  Interventions: Device: GE OPTIMA MR430s with HDX/GE Electronics

INTERVENTIONS:
Device: GE OPTIMA MR430s with HDX/GE Electronics — MRI scan(s) for no longer than 60 minutes

SUMMARY:
The purpose of this study is to determine the safety of a customized MRI scanner and gather preliminary data on image quality in a group of 10 medically stable infants admitted to the Neonatal Intensive Care Unit (NICU) at Cincinnati Children's Hospital Medical Center (CCHMC).

DETAILED DESCRIPTION:
The current practice of transferring infants from the Neonatal Intensive Care Unit (NICU) to radiology departments and imaging in adult-sized magnetic resonance imaging (MRI) scanners is associated with significant safety and image quality issues. For these reasons, the potential of MRI for diagnosing disease in neonates has yet to be fully realized. The overreaching goal of our research effort is to bring high-performance MRI into the NICU so that neonates can benefit from the same quality of diagnostic imaging as adults. To accomplish this we have converted a commercial small-bore 1.5 Tesla (T) MRI scanner designed for orthopedic use into a neonatal MRI system optimized for whole body imaging of neonates. The purpose of this initial study is to determine the safety of the customized scanner installed in the NICU at Cincinnati Children's Hospital Medical Center (CCHMC) and gather preliminary data on image quality in a group of 10 medically stable infants admitted to the CCHMC NICU.

ELIGIBILITY:
Inclusion Criteria:

* Any infant admitted to the NICU at CCHMC
* Medically stable as per the opinion of the attending neonatologist currently on service
* Parental consent obtained

Exclusion Criteria:

* Infants too large to fit in the customized NICU MRI system comfortably (expected to be infants >4.5 kg)
* Standard MRI exclusion criteria as set forth by the CCHMC Division of Radiology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Dumoulin, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- NICU, Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients, eligible to participate, were recruited from within the NICU beginning in February 2012 ending in April 2012.
Pre-assignment Details: All participants enrolled in the study, completed the study.
Groups:
- Pilot Group: Patients who received an MRI.
Period: Overall Study
Arm/Group | Pilot Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot Group: Patients who had an MRI in the NICU scanner.
Arm/Group | Pilot Group
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | .19 (.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as Measured by Vital Signs, Change in Temperature, and Physical Exam
Description: Heart rate and oxygen saturation will be measured every 15+/- 5 minutes. The infants' temperatures will be taken immediately before the MRI and again immediately after the MRI. A physical exam will be performed both immediately before and immediately after the MRI to assess for any physical changes.
Time Frame: Day 1
Measure: Number; unit: Adverse Events
Groups:
- Pilot Group: Patients who received an MRI on the NICU scanner.
Arm/Group | Pilot Group
Number analyzed (Participants) | 15
Adverse Events | 0

2. Secondary Outcome: MRI Image Quality
Description: The following measures will be individually evaluated and compared to similar images previously acquired on an adult scanner: Overall Study Quality, Motion, Spatial Resolution, Signal to Noise, and Contrast.
Time Frame: Post MRI Scan for Each Infant
Population: Number of NICU MRI Images with Equal or Better Quality than Adult Scanner Images
Measure: Number; unit: Images
Groups:
- Pilot Group: Patients who had an MRI on the NICU scanner.
Arm/Group | Pilot Group
Number analyzed (Participants) | 15
Images | 15

ADVERSE EVENTS:
Time Frame: Patients were monitored for approximately 2 hours after the MRI for Adverse Events for skin changes due to the monitor leads.
Description: Patients' vital signs (heart rate and oxygen saturation) were measured and recorded during the MRI. The physician present performed a physical exam immediately after the MRI to assess for any skin changes due to the MRI scan process.
Arm/Group | Pilot Group
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Group (N=15)
Mild Desaturation (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Baby had a mild desaturation for about 5 seconds. It was unrelated to the study.
Drop in Heart Rate (Cardiac disorders) | 1 (1) — One baby had a drop in heart rate for about 5 seconds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No